CLINICAL TRIAL: NCT03860714
Title: Correlation Between Urine UACR and Postoperative Neurocognitive Disorder in Elderly Patients With Non-cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Han Yuan (Other)
Responsible Party: Sponsor-Investigator, Han Yuan, Doctor-in-charge of Anesthetist, Xuzhou Medical University
Organization: Xuzhou Medical University (Other)
Other Study IDs: XYFY2019-KL015-01
Record Dates: First submitted 2019-02-22; First posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Cognitive Dysfunction; Delirium
Keywords: Postoperative Cognitive Dysfunction; Delirium; UACR
MeSH Terms: conditions — Postoperative Cognitive Complications; Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — urine and blood

GROUPS / COHORTS (1):
- study group: 400 Male and female patients undergoing non-cardiac surgery at the Affiliated Hospital of Xuzhou Medical University [Jiangsu China].We do the neuropsychological tests,MMSE,CCI，CDR,QoR-40,GDS,CAGE Alcoholism Questionnaire，Pure Tone Audiometry，blood albumin、hemoglobin content、ALT、AST、BUN、Cr、serum folic acid、vitamin B12、homocysteine and branched chain amino acid content 1 day before the surgery（baseline）； 1 day before the surgery（baseline）； Confusion Assessment Method（CAM)，NRS once before discharge from PACU and 1、2、3 days after surgery twice a day； QoR-40 1 day after surgery； Neuropsychological tests and MMSE 6±1 days and one month after surgery.
  Interventions: Diagnostic Test: Neuropsychological tests

INTERVENTIONS:
Diagnostic Test: Neuropsychological tests — We do the neuropsychological tests, Mini-Mental score examination (MMSE),Charlson Comorbidity Index(CCI)，Clinical Dementia Rating(CDR),Quality of Recovery Score - 40 (QoR-40),Geriatric Depression Scale (GDS),CAGE Alcoholism Questionnaire，Pure Tone Audiometry，blood albumin、hemoglobin content、ALT、AST、BUN、Cr、serum folic acid、vitamin B12、homocysteine and branched chain amino acid content 1 day before the surgery（baseline）； 1 day before the surgery（baseline）； Confusion Assessment Method（CAM)，Numerical Rating Scale（NRS）once before discharge from PACU and 1、2、3 days after surgery twice a day； QoR-40 1 day after surgery； Neuropsychological tests and MMSE 6±1 days and one month after surgery.

SUMMARY:
This study intends to evaluate the relationship between urinary albumin/creatinine ratio and postoperative neurocognitive impairment in elderly non-cardiac surgery patients. The results of the study are to identify risk factors, screen high-risk populations to improve clinical evidence, early detection and early treatment.And reducing the burden of PNCD on patients and their families, hospitals and public resources.

ELIGIBILITY:
Inclusion Criteria:

* Non-cardiac surgery patients;

  * Age is greater than or equal to 60 years old; ③Han Nationality, mother tongue is chinese;

    ④The MMSE score:Illiteracy is greater than or equal to 17 points, primary school is greater than or equal to 20 points, higher secondary school is more than 24 points;

    ⑤The people signed informed consent.

Exclusion Criteria:

* The diagnosis of preoperative delirium；

  * The diagnosis Unstable hypertension（Such as：pheochromocytoma or aortic dissection）； ③Severe chronic obstructive pulmonary disease or congestive heart failure； ④Severe liver and kidney dysfunction;

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included 400 patients undergoing non-cardiac surgery at the affiliated hospital of Xuzhou Medical University.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Confusion Assessment Method（CAM) | before discharge from PACU
  Confusion Assessment Method to measure delirium
Confusion Assessment Method（CAM) | morning of the 1st day after surgery
  Confusion Assessment Method to measure delirium
Confusion Assessment Method（CAM) | afternoon of the 1st day after surgery
  Confusion Assessment Method to measure delirium
Confusion Assessment Method（CAM) | morning of the 2st day after surgery
  Confusion Assessment Method to measure delirium
Confusion Assessment Method（CAM) | afternoon of the 2st day after surgery
  Confusion Assessment Method to measure delirium
Confusion Assessment Method（CAM) | morning of the 3st day after surgery
  Confusion Assessment Method to measure delirium
Confusion Assessment Method（CAM) | afternoon of the 3st day after surgery
  Confusion Assessment Method to measure delirium

SECONDARY OUTCOMES:
Quality of Recovery Score - 40 (QoR-40) | 1 day before surgery(baseline)
  Quality of recovery will be evaluated by Quality of Recovery 40 (QoR40),which assesses five dimensions of recovery (physical comfort,emotional state, physical independence , physiological support and pain ). Each item is rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery).
Quality of Recovery Score - 40 (QoR-40) | 1 day after surgery
  Quality of recovery will be evaluated by Quality of Recovery 40 (QoR40),which assesses five dimensions of recovery (physical comfort,emotional state, physical independence , physiological support and pain ). Each item is rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery).
Numerical Rating Scale（NRS） | before discharge from PACU
  Evaluate the severity using numerical rating scale（NRS）, where zero mean no pain and 10 the worst imaginable pain.
Numerical Rating Scale（NRS） | morning of the 1st day after surgery
  Evaluate the severity using numerical rating scale（NRS）, where zero mean no pain and 10 the worst imaginable pain.
Numerical Rating Scale（NRS） | afternoon of the 1st day after surgery
  Evaluate the severity using numerical rating scale（NRS）, where zero mean no pain and 10 the worst imaginable pain.
Numerical Rating Scale（NRS） | morning of the 2st day after surgery
  Evaluate the severity using numerical rating scale（NRS）, where zero mean no pain and 10 the worst imaginable pain.
Numerical Rating Scale（NRS） | afternoon of the 2st day after surgery
  Evaluate the severity using numerical rating scale（NRS）, where zero mean no pain and 10 the worst imaginable pain.
Numerical Rating Scale（NRS） | morning of the 3st day after surgery
  Evaluate the severity using numerical rating scale（NRS）, where zero mean no pain and 10 the worst imaginable pain.
Numerical Rating Scale（NRS） | afternoon of the 3st day after surgery
  Evaluate the severity using numerical rating scale（NRS）, where zero mean no pain and 10 the worst imaginable pain.
Mini-Mental score examination (MMSE) | 1 day before surgery(baseline)
  Mini-Mental score examination [MMSE] used for screening of dementia
Mini-Mental score examination (MMSE) and Neuropsychological tests | 6±1 days after surgery
  Mini-Mental score examination (MMSE) and Neuropsychological tests to measure cognitive function, including the Trail
Mini-Mental score examination (MMSE) and Neuropsychological tests | one month after surgery
  Mini-Mental score examination (MMSE) and Neuropsychological tests to measure cognitive function, including the Trail
serum folic acid levels | 1 day before surgery(baseline)
  Record preoperative serum folic acid levels
serum vitamin B12 levels | 1 day before surgery(baseline)
  Record preoperative serum vitamin B12 levels
serum homocysteine content | 1 day before surgery(baseline)
  Record preoperative serum homocysteine content
serum branched chain amino acid content | 1 day before surgery(baseline)
  Record preoperative serum branched chain amino acid content

OTHER OUTCOMES:
blood Albumin levels | before surgery(baseline)
  Record preoperative blood Albumin levels
blood Hemoglobin content | before surgery(baseline)
  Record preoperative blood Hemoglobin content
blood Alanine aminotransferase （ALT） levels | before surgery(baseline)
  Record preoperative blood Alanine aminotransferase （ALT） levels
blood Aspartate aminotransferase （AST）levels | before surgery(baseline)
  Record preoperative blood Aspartate aminotransferase （AST）levels
Blood urea nitrogen（BUN） levels | before surgery(baseline)
  Record preoperative Blood urea nitrogen（BUN） levels
Blood creatinine（Cr） levels | before surgery(baseline)
  Record preoperative Blood creatinine（Cr） levels

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia of the Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China